CLINICAL TRIAL: NCT01174654
Title: Development of a Methamphetamine Early Intervention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21DA019420-01A1 (NIH); R21DA019420-01A1 (NIH)
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: HIV; Sexual Behavior; Methamphetamine; Behavioral Research
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Referral to community resources (No Intervention)
- Contingency Management (Experimental)
  Interventions: Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Contingency management — A 12-week contingency management intervention
  Other Names: Voucher-based reinforcement
  Arms: Contingency Management

SUMMARY:
Methamphetamine abuse has a strong and consistent epidemiologic association with high-risk sexual behavior and both prevalent and incident HIV in men who have sex with men (MSM), and some authorities have advocated methamphetamine treatment as an HIV prevention strategy. However, methamphetamine interventions have not been evaluated in controlled trials, nor have they been implemented and assessed outside of substance abuse treatment programs. This application proposes preliminary investigations to adapt a methamphetamine treatment intervention previously associated with decreased sexual-risk taking among MSM for use as an early intervention among MSM in Seattle, Washington. Sixty methamphetamine-using MSM will be enrolled in a randomized controlled trial of contingency management (CM) versus no intervention. CM participants will have their urine tested for methamphetamine 3 times weekly for 12 weeks, and will receive vouchers of escalating value when their urines test negative; vouchers will be withheld when participants' urines test positive for methamphetamine or participants miss urine testing visits. All participants will undergo urine methamphetamine testing and audio-computer assisted self-interviews on sexual behavior and substance use at baseline and at 6 week intervals for 6 months. Participants will be tested for HIV, syphilis, rectal gonorrhea and chlamydial infection, and pharyngeal gonorrhea at baseline and at 3 and 6 month follow-up. The study will determine how often MSM will initiate and complete the early intervention, and will longitudinally measure unsafe sexual behaviors among intervention and control participants. Study results will determine the feasibility of instituting and studying CM as an early intervention; define whether the intervention is sufficiently promising to justify a larger, definitive randomized controlled trial; and will provide estimates for defining the number of participants such a trial would require.

ELIGIBILITY:
Inclusion Criteria:

* Anal sex with another man in the month prior to enrollment
* Use of methamphetamine on at least 2 days in the month prior to enrollment

Exclusion Criteria:

* Plans to move from the study catchment area within 6 months of enrollment
* A mutually monogamous relationships with a man of the same HIV status lasting 2 or more years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Non-concordant unprotected anal intercourse | Baseline, 6, 12, 18, 24 weeks

SECONDARY OUTCOMES:
Number of non-concordant unprotected anal intercourse partners | Baseline, 6, 12, 18, 24 weeks
Stimulant (methamphetamine and crack/cocaine) urinalyses | Baseline, 6, 12, 18, 24 weeks
Self-reported methamphetamine use | Baseline, 6, 12, 18, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Golden, Principal Investigator — University of Washington
Locations (1):
- Lifelong AIDS Alliance, Seattle, Washington, United States

REFERENCES:
- [Derived] Menza TW, Jameson DR, Hughes JP, Colfax GN, Shoptaw S, Golden MR. Contingency management to reduce methamphetamine use and sexual risk among men who have sex with men: a randomized controlled trial. BMC Public Health. 2010 Dec 20;10:774. doi: 10.1186/1471-2458-10-774. PMID 21172026